CLINICAL TRIAL: NCT01481753
Title: Pancreaticoduodenectomy With or Without Braun Enteroenterostomy: Comparison of Postoperative Pancreatic Fistula and Delayed Gastric Emptying
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: last patient recruited Feb 2015,completion of data review; study data do not meet statistical significance to answer proposed study question
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00021168
Record Dates: First submitted 2011-11-10; First posted 2011-11-30 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Pancreatic Fistula; Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Braun arm (Active Comparator): patients received Braun enteroenterostomy
  Interventions: Procedure: Braun enteroenterostomy
- Non Braun Arm (Active Comparator): Patients do not receive a Braun enteroenterostomy
  Interventions: Procedure: pancreaticoduodenectomy without Braun enteroenterostomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy without Braun enteroenterostomy — no Braun enteroenterostomy has been added to standard pancreaticoduodenectomy; pancreaticoduodenectomy without Braun enteroenterostomy
  Other Names: No Braun
  Arms: Non Braun Arm
Procedure: Braun enteroenterostomy — addition of Braun enteroenterostomy (side-to-side anastomosis between the afferent and efferent loops of the gastrojejunostomy) to standard PD reconstruction can decrease the rates of POPF and/or DGE, improving the perioperative outcome of patients undergoing PD.
  Arms: Braun arm

SUMMARY:
The investigators plan to perform a prospective randomized, head-to-head trial to test the hypothesis that the addition of Braun enteroenterostomy to standard pancreaticoduodenectomy (PD) reconstruction can decrease the rates of Postoperative Pancreatic Fistula (POPF) and/or Delayed Gastric Emptying (DGE).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy surgery at Johns Hopkins Hospital

Exclusion Criteria:

* Pregnant women
* Patients under the age of 18
* adults lacking ability to consent,
* patients scheduled for laparoscopic whipple surgery
* non-english-speakers, and
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2009-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Decreased rates of pancreatic fistula in surgeries adding Braun enteroenterostomy | patients will be followed during hospital stay and interviewed at 90 days +/- 2 weeks post surgery
  patients will be assessed for post operative fistula and delayed gastric emptying during hospitalization and then interviewed at 90 days +/- 2 weeks from OR date to assess any unanticipated consequences after discharge. We are currently performing statistical analysis of outcome data on the first 100 consented whipple patients as outlined in Johns Hopkins Hospital (JHH)-approved Institutional Review Board (IRB) protocol.

SECONDARY OUTCOMES:
Reduced incidence of delayed gastric emptying in patients with Braun enteroenterostomy | patients will be followed during hospital stay and interviewed at 90 days +/- 2 weeks post surgery
  patients will be assessed for post operative fistula and delayed gastric emptying during hospitalization and then interviewed at 90 days +/- 2 weeks from OR date to assess any unanticipated consequences after discharge We are currently performing statistical analysis of outcome data on the first 100 consented whipple patients as outlined in JHH-approved IRB protocol

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Wolfgang, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States